CLINICAL TRIAL: NCT05890430
Title: Study of Alloimmune Response in Humoral Rejection After Kidney Transplantation "REjet Cellules Immunitaires Transplantation rEnale" (RECITE)
Brief Title: Study of Alloimmune Response in Humoral Rejection After Kidney Transplantation
Acronym: RECITE
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 8968
Record Dates: First submitted 2023-05-25; First posted 2023-06-06 (Actual); Last update posted 2023-06-08 (Actual); Status verified 2023-05

CONDITIONS: Kidney Transplantation; Kidney Allograft Biopsy; Humoral Rejection; Microvascular Inflammation
Keywords: Kidney Transplantation; Humoral rejection; Kidney allograft biopsy; Alloimmunization; Genetic incompatibilities
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood Urine Graft biopsies
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with microvascular inflammation: Patients presenting with microvascular inflammation on kidney allograft biopsy
  Interventions: Biological: Blood draw, Urine draw
- Patient without microvascular inflammation: Patients presenting without microvascular inflammation on kidney allograft biopsy
  Interventions: Biological: Blood draw, Urine draw

INTERVENTIONS:
Biological: Blood draw, Urine draw — Collection of an additional volume of blood at each follow-up time in addition to the standard blood test performed during the patient's follow-up Collection of an additional volume of urine at each follow-up time

SUMMARY:
We will study a prospective cohort including all kidney transplant recipients undergoing kidney graft biopsy in one kidney transplantation center, for a duration of 5 years.

Our primary outcome is to compare the number of circulating NK cells between patients and without humoral rejection.

Our secondary outcomes are to describe the cellular, genetic, humoral, and histological characteristics of humoral rejection and their evolution.

DETAILED DESCRIPTION:
Information and inclusion visit (V0) The information and inclusion visit will be carried out on the day of the graft biopsy or, in the case of pre-scheduled biopsies, during a consultation prior to the biopsy (still as part of standard follow-up). This is particularly the case for patients undergoing systematic biopsy. The indication for graft puncture-biopsy is generally decided by the nephrologist in charge of the patient, or at departmental meetings for complex cases.

During this consultation, the physician verifies the inclusion criteria and obtains the patient's consent to take part in the study. We explain to the patient the scientific interest of evaluating the immune response in humoral rejection, and the absence of repercussions for the patient's subsequent management. A routine clinical examination is performed, and the patient's current treatment regimen is notified.

If the patient agrees, a blood sample is taken for the standard biology follow-up of transplant patients and for the study samples:

* Serum factors: 4 dry tubes or SST or EDTA 5 ml maximum
* PBMCs: 8 heparinized tubes of 10 ml maximum, which may be replaced by Paxgen tubes in case of technical or logistical necessity
* Urine: 5 dry tubes or SST 5 ml maximum

Patients will be divided into two groups according to the indication for biopsy, with an influence on follow-up:

* patients who underwent systematic biopsy (M3 and M12)
* patients included in a biopsy for cause, whatever the distance to the graft

Follow-up visits (V1, V2, V3, etc.) Subsequently, new samples may be offered to included patients, in order to compare the parameters studied at the time of and after their graft biopsies. The different follow-up times are indexed to the standard follow-up of kidney transplant patients.

-Patients routinely biopsied between M0 and M6 of transplantation (most often M3): Follow-up will be indexed to post-transplant consultation follow-up. New samples may be taken at M6, M9, M12 (at the time of the second systematic biopsy), M18, M24 of transplantation or during a follow-up biopsy.

Patients biopsied for cause, at any time post-transplant: follow-up will be indexed to the completion of patient follow-up consultations. New samples may be taken at M3, M6, M9, M12, M18, M24 after the biopsy, or during a follow-up biopsy.

With the patient's consent, blood and urine samples are taken for the standard follow-up biology of transplant patients and for the study samples:

* Serum factors: 4 dry tubes or SST or EDTA 5 ml maximum
* PBMCs: 8 heparinized tubes of 10 ml maximum, which may be replaced by Paxgen tubes in case of technical or logistical necessity
* Urines: 5 dry tubes or SST 5 ml

ELIGIBILITY:
Inclusion Criteria:

* Kidney transplant recipient, male or female, 18 years of age or older
* Patient undergoing a kidney allograft biopsy, according to the usual protocol of the service
* Subject affiliated with a social health insurance scheme.
* Subject capable of understanding the objectives and risks associated with the research and expressing non-opposition

Exclusion Criteria:

* Inability to provide the subject with clear and proper information (difficulties in understanding the subject, ...)
* Refusal of the patient to participate in the study
* Subject under guardianship or curatorship
* Subjects under legal protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All kidney transplant recipients undergoing a kidney allograft biopsy for a duration of five years in a single kidney transplantation center.
Sampling Method: Non-Probability Sample
Enrollment: 570 (Estimated)
Dates: Start 2023-06 (Estimated); Primary Completion 2033-06 (Estimated); Study Completion 2033-07 (Estimated)

PRIMARY OUTCOMES:
Number of circulating CD3- CD56+ cells | Day of inclusion sample (= day of kidney allograft biopsy)
  Comparison between patients with microvascular inflammation and other patients